CLINICAL TRIAL: NCT04606355
Title: Autostereoscopic Dynamic Near Vision Testing of Acuity, Stereo and Color on PDI Check
Brief Title: Autostereoscopic Dynamic Near Vision Testing
Acronym: PDICheck
Status: Suspended | Type: Observational
Why Stopped: updated technology nearly ready
Sponsor: Alaska Blind Child Discovery (Other)
Responsible Party: Sponsor
Other Study IDs: PDICheck
Record Dates: First submitted 2020-10-22; First posted 2020-10-28 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Visual Suppression; Amblyopia; Color Vision Defects
Keywords: stereopsis, visual acuity
MeSH Terms: conditions — Amblyopia; Color Vision Defects | interventions — Visual Acuity; Color Vision

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PDI Check & Conventional: Autostereoscopic, dynamic forced choice game (ie on Nintendo 3DS) and Rosenbaum or HOTV near card, Ishihara color plates, Innova Rabin color test, Titmus Stereo test
  Interventions: Diagnostic Test: Visual Acuity; Diagnostic Test: stereopsis; Diagnostic Test: Color vision

INTERVENTIONS:
Diagnostic Test: Visual Acuity — autostereoscopic, monocular dynamic force choice test
Diagnostic Test: stereopsis — autostereoscopic dynamic forced-choice depth perception test
Diagnostic Test: Color vision — autostereoscopic forced choice monocular or binocular color vision tests

SUMMARY:
This is an analysis of tests of near vision.

Visual perception testing using a novel program on an interactive three dimensional electronic device:

Autostereoscopic dynamic near games for monocular visual acuity, stereopsis and color are compared with other conventional or similar tests.

DETAILED DESCRIPTION:
Subjects with normal vision, exceptional vision, or visual deficits have near vision tested on the PDI Check game and compared to other clinical tests.

Interclass Correlation and Bland Altman analysis utilized for continuous data. Sensitivity and Specificity calculated for defined clinical entities. Subjects are not assigned to either one screening test or another; instead different tests are compared.

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects, patients with deficient binocular vision, patients with color vision disorders

Exclusion Criteria:

* phthisis, enucleations

Ages: 1 Year to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Normal subjects and patients with near vision disorders
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-11-16 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity | day 1
  Gold Standard clinical test of visual acuity
stereopsis | day 1
  Gold standard clinical test of stereopsis (ie Titmus)
Color Vision | day 1
  Gold Standard clinical test of color vision (Ishihara, Innova Rabin)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle A Smith, OD, Principal Investigator — Alaska Blind Child Discovery
Locations (1):
- Alaska Blind Child Discovery, Anchorage, Alaska, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified database on www.ABCD-Vision.org
Time Frame: 1 year after recruitment, then ongoing
Access Criteria: de-identified to any investigator with web access
URL: http://www.abcd-vision.org/references/index.html

REFERENCES:
- [Background] Smith KA, Arnold AW, Sprano JH, Arnold SL, Arnold RW. Performance of a Quick Screening Version of the Nintendo 3DS PDI Check Game in Patients With Ocular Suppression. J Pediatr Ophthalmol Strabismus. 2019 Jul 1;56(4):234-237. doi: 10.3928/01913913-20190502-01. PMID 31322713
- [Background] Martin SJ, Rowe KS, Hser N, Htoo HE, Khin R, Smith KA, Arnold RW. Compared Near-Vision Testing With the Nintendo 3DS PDI Check Game on the Thai-Burma Border. Asia Pac J Ophthalmol (Phila). 2019 Jul-Aug;8(4):330-334. doi: 10.1097/APO.0000000000000251. PMID 31385820
- [Background] Smith KA, Damarjian AG, Molina A, Arnold RW. Calibrated measurement of acuity, color and stereopsis on a Nintendo(R) 3DS game console. Clin Optom (Auckl). 2019 Apr 30;11:47-55. doi: 10.2147/OPTO.S199992. eCollection 2019. PMID 31118854
- [Background] Vancleef K, Serrano-Pedraza I, Sharp C, Slack G, Black C, Casanova T, Hugill J, Rafiq S, Burridge J, Puyat V, Enongue JE, Gale H, Akotei H, Collier Z, Haggerty H, Smart K, Powell C, Taylor K, Clarke MP, Morgan G, Read JCA. ASTEROID: A New Clinical Stereotest on an Autostereo 3D Tablet. Transl Vis Sci Technol. 2019 Feb 28;8(1):25. doi: 10.1167/tvst.8.1.25. eCollection 2019 Jan. PMID 30834173
- [Background] Fanlo Zarazaga A, Gutierrez Vasquez J, Pueyo Royo V. Review of the main colour vision clinical assessment tests. Arch Soc Esp Oftalmol (Engl Ed). 2019 Jan;94(1):25-32. doi: 10.1016/j.oftal.2018.08.006. Epub 2018 Oct 22. English, Spanish. PMID 30361001
- [Background] Arnold R, Angi M. Multifaceted Amblyopia Screening with blinq, 2WIN, and PDI Check. Clin Ophthalmol. 2022 Feb 15;16:411-421. doi: 10.2147/OPTH.S349638. eCollection 2022. PMID 35210746
- [Background] Mahlen T, Arnold RW. Pediatric Non-Refractive Vision Screening with EyeSwift, PDI Check and Blinq: Non-Refractive Vision Screening with Two Binocular Video Games and Birefringent Scanning. Clin Ophthalmol. 2022 Feb 11;16:375-384. doi: 10.2147/OPTH.S344751. eCollection 2022. PMID 35177896
- [Background] Brown S, Rue C, Smith K, Arnold R. Extraordinary Dynamic Near Vision in Champion Shotgun Shooters: PDI Check Evaluation of Stereo and Color without Floor Effect. Clin Ophthalmol. 2021 Feb 16;15:575-581. doi: 10.2147/OPTH.S298234. eCollection 2021. PMID 33623358
- [Background] Arnold A, Smith K, Molina A, Damarjian A, Desatoff T, Arnold R. Trichromatic Enhanced Dynamic Color Screening on the PDI Check Nintendo 3DS Game. Clin Optom (Auckl). 2021 May 11;13:137-141. doi: 10.2147/OPTO.S305042. eCollection 2021. PMID 34007233
- See also: device website — http://www.pdicheck.com